CLINICAL TRIAL: NCT03589352
Title: Women's Knowledges About Gynaecological Aftercare, Hospitalized in Maternity Service, or Consulting in Policlinic, in University Hospitals of Strasbourg
Brief Title: Women's Knowledges About Gynaecological Aftercare
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7101
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Gynecology
Keywords: gynaecological aftercare; contraception; breast cancer; cervix cancer; cervical screening; breast self examination; mammography; midwife; body knowledge; prevention; self care
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Breast Self-Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hypothesis of the investigators is that women don't have all the needfull knowledge to understand the importance of a regular gynaecological aftercare.

The main objective is to assess women's knowledge's about gynaecological aftercare.

The second objective is to identify barriers that prevent women of a regular gynaecological aftercare

ELIGIBILITY:
Inclusion Criteria:

* women aged over eighteen years old
* women who are able to read and write French

Exclusion Criteria:

* women aged under eighteen years old
* women who aren't able to read or write French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - women who are able to read and write French
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
questionnaire | 24 hours before the discharge of patients from the gynecology department
  Assessment of women's knowledge of gynecological follow-up via a questionnaire. The score is calculated from the questionnaire 24 hours before the discharge of patients from the gynecology department

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie (CMCO), Strasbourg, France